CLINICAL TRIAL: NCT04078113
Title: Stimulation Anda Validation of the Pupillary Dilation for the Detection of Pain in Analgosedated Patients Under Mechanically in Intensive Care Unit
Brief Title: Stimulation and Validation of the Pupillary Dilation for the Detection of Pain in Analgosedated Patients Under Mechanically Ventilation in Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Ana Vallejo de la Cueva, Principal Investigator, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PUPIPAIN
Record Dates: First submitted 2019-07-02; First posted 2019-09-04 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Pain
Keywords: Pupillary dilation; Analgosedated; Mechanically ventilation
MeSH Terms: conditions — Pain; Mydriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Every patient will be subjected to a measured stimulus with a power selected in phase 1 (X mA) and pupillary dilatation will be measured by pupillometry. In those patients showing pupillary size variation over the limit for insufficient analgesia estimated in phase 1 for tracheal suction, additional analgesia will be provided before tracheal suction. In those patients without pain detected by pupillometry, additional anlagesia won´t be provided. In both cases Pupillometry, BPS and ESCID will be measured during tracheal suction to determine whether the patient is in pain or not.
  Interventions: Other: Pupillometer
- Control group (No Intervention): Before tracheal suction and due to medical decision, analgesia following current clinical practice would be administered prophylactically.
  Pupillometry, BPS and ESCID will be measured during tracheal suction to determinate whether the patient is in pain or not.

INTERVENTIONS:
Other: Pupillometer — Measurements of pupillary dilatation with pupillometer to administer or not analgesia
  Arms: Experimental group

SUMMARY:
This project has 2 phases. Phase 1: diagnostic test study, to evaluate the efficacy of the variation of pupillary size (PDR) to detect pain in ICU patients regarding to Behavioural Pain Scale (BPS) and ESCID (Conductual Scale Pain Index). Phase 2: controlled and aleatorized clinical trial to evaluate efficacy in PDR monitoring after painful assessed minimum stimulus with the best diagnostic efficiency on phase 1, as a need of analgesia indicator tool.

The sample will be patients over 18 years, sedated and mechanically ventilated, with an initial BPS of 3, RASS between -1 and -4, not able not to communicate , with inform consent signed. Exclusion criteria will be: ophtalmologic pathology and administration of drugs interfering pupillary reflexes. Measurements before/during pain/non-pain situations, aspiration of secretions and calibrated intensity stimulus through the pupilometer Algiscan. The investigators will study association between pain according to BPS/ESCID and pupillary dilatation according to pupillometry and percentage of patients with pain and preanalgesia according to pupillometry and standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years.
* Analgosedated patients under mechanical ventilation.
* Unable to communicate (verbal or motor).
* Patients with initial BPS of 3, and RASS from -1 to -4.
* Familiar prior informed consent.

Exclusion Criteria:

* Patients treated with muscle relaxants.
* Severe Critical Polyneuropathy.
* Pupillary reflex affectation in diabetic patients (diabetic papillopathy,glaucomatous optic neuropathy) or any other pathologies like Adie´s Syndrome, Argyl-Robertson pupil.
* Patients with tansmisible ocular infections.
* Patients with possible injury of the third carnial nerve (Horner´s syndrome) due to injury to the brainstem, cervical cord, cancer of the upper lobe the lung, dissection of the carotid and/or cluster headache.
* Acute cerbrovascular conditions with Glasgow Coma Scale less than 6, or increased intracranial pressure, or pontine base infarction.
* Drugs that interfere with the pupillary reflex (clonidine, dexmedetomidine, metoclopramide, tramadol, droperidol, ketamine, nitrous oxide).
* Patients under metoclopramide, if given 10 minutes prior the measurement of the pupillary reflex (PDR).
* Patients during the first 24 hours after Cardiac Arrest (CRP).
* Severe unestable comorbidity with doses of norepinephrine> 0.6 microg/kg/min and/or dobutamine>10 microg/kg/min or drenalin any doses.
* Patients with untreated pheochromocytomas.
* Refuse to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Propotion of patient with pain on experimental group versus control group | An average of 1 year
  To compare the proprtion of patients with pain according to Behavioral Pain Scale (BPS), pupillometry and Scale of Behaviour Indicators of Pain (escid)
Proportion of patient who require anesthesia on experimental group versus control group | An average of 1 year
  The proportion of patients who require anesthesia on experimental group (previous analgesia according to pupillometry during endotracheal aspiration) versus control group (previous analgesia according to standard clinical practice).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Vallejo de la Cueva, Dr., Principal Investigator — Basque Health System
Locations (1):
- Araba University hospital, Vitoria-Gasteiz, Álava, Spain

REFERENCES:
- [Derived] Lopez de Audicana Jimenez de Aberasturi Y, Vallejo De la Cueva A, Parraza Diez N. The effectiveness of a pupillary dilation reflex as an analgesia indicator: A protocol for a randomised multicentre trial in critically ill patients. Int J Nurs Stud Adv. 2025 Oct 1;9:100431. doi: 10.1016/j.ijnsa.2025.100431. eCollection 2025 Dec. PMID 41159095
- [Derived] Lopez-De-Audicana-Jimenez-De-Aberasturi Y, Vallejo-De-La-Cueva A, Parraza-Diez N. Behavioral pain scales, vital signs, and pupilometry to pain assessment in the critically ill patient: A cross sectional study. Clin Neurol Neurosurg. 2024 Dec;247:108644. doi: 10.1016/j.clineuro.2024.108644. Epub 2024 Nov 18. PMID 39571502
- [Derived] Lopez de Audicana-Jimenez de Aberasturi Y, Vallejo-De la Cueva A, Aretxabala-Cortajarena N, Rodriguez-Nunez C, Pelegrin-Gaspar PM, Gil-Garcia ZI, Rodriguez-Borrajo MJ, Marguello-Fernandez AA, Parraza-Diez N. The pupillary dilation reflex to a nociceptive stimulus as a tool for analgesia management: A diagnostic study. Aust Crit Care. 2024 Mar;37(2):230-235. doi: 10.1016/j.aucc.2023.06.009. Epub 2023 Aug 10. PMID 37573155